CLINICAL TRIAL: NCT02610660
Title: Tracking Outcomes and Practice in Pediatric Pulmonary Hypertension
Acronym: TOPP-2
Status: Completed | Type: Observational
Sponsor: Association for Pediatric Pulmonary Hypertension (Other)
Responsible Party: Sponsor
Other Study IDs: TOPP-2
Record Dates: First submitted 2015-11-10; First posted 2015-11-20 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The TOPP-2 registry is an international, non-interventional, prospective registry including children and adolescents newly diagnosed with pulmonary hypertension (PH) to gain further insights in the disease course and long-term outcome of PH in childhood.

Patients will undergo clinical assessments and receive standard medical care, as determined by treating physicians in their daily clinical practice. The TOPP-2 registry is specifically designed to capture the variables that have been proposed as treatment goals in PePH and the reasons for changes in treatment strategy.

The TOPP-2 registry uses the new clinical classification of PH as outlined at the 5th World Symposium for Pulmonary Hypertension (WSPH) in Nice 2013 and includes new characterizations for children with PH.

The registry is planned and implemented under the scientific leadership of the Association for Pediatric Pulmonary Hypertension (PePH), independently from the financial sponsors.

All enrolled patients will have a follow-up period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be an incident patient, i.e.newly diagnosed with PH
* Age at time of diagnosis is at least 3 months and less than 18 years
* Patients must present with PH belonging to one of the following categories

  * Group 1 according to updated Nice clinical classification
  * Group 3 according to updated Nice clinical classification
  * Group 4 according to updated Nice clinical classification
  * Group 5 according to updated Nice clinical classification
* PH confirmed by heart catheterisation (HC)
* At HC, the patient must present with mean pulmonary arterial pressure (PAP) of at least 25 mmHg at rest, a pulmonary vascular resistance index (PVRi) equal to or below 3 Wood units*m^2 and mean pulmonary arterial wedge pressure (PAWP) below or equal to 15 mmHg
* In case of congenital heart disease (CHD) patients who had undergone palliative procedure or repair to close systemic to pulmonary shunt, the diagnosis of PH must have been confirmed by HC at least 6 months after surgery/palliative procedure took place
* For patients with PAH-CHD open shunt, only those considered not operable due to advanced pulmonary vascular disease are eligible
* Patients to be included into the registry, and/or their legal guardians, must give informed consent. Where applicable patients will be asked for their written assent
* Participating sites must agree to adhere to the recommendations of the WSPH 2015 Nice, Pediatric Taskforce.

Exclusion Criteria:

* Patients belonging to Group 2 according to updated Nice clinical classification

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Children and adolescents, newly diagnosed with PH (incident PePH patients), meeting the inclusion criteria. A patient is considered an incident patient if the time elapsed between the diagnostic RHC and the initial visit at the site including the patient is less than or equal to three months and if the time between diagnostic RHC and informed consent is less than or equal to six months
  2. Ex-incident patients from the previous TOPP-1 registry.
Sampling Method: Non-Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2015-08; Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Death | Over registry run-time (5.5 years)
Transplantation | Over registry run-time (5.5 years)
Adverse events | Over registry run-time (5.5 years)

SECONDARY OUTCOMES:
Hospitalisation related to pulmonary arterial hypertension (PAH) | Over registry run-time (5.5 years)
Use/initiation of i.v./s.c. prostanoids | Over registry run-time (5.5 years)
Atrial septostomy | Over registry run-time (5.5 years)
Potts shunt | Over registry run-time (5.5 years)
Time to clinical worsening | Over registry run-time (5.5 years)
  Various composites of above parameters
Decline in 6-minute walk test (6MWT) | Over registry run-time (5.5 years)
Type of treatment | Over registry run-time (5.5 years)
  Type of treatment (drug, mono/combination, administration route)
Switch in treatment | Over registry run-time (5.5 years)
Escalation of treatment | Over registry run-time (5.5 years)
Reasons for treatment change | Over registry run-time (5.5 years)
Decline in WHO functional class | Over registry run-time (5.5 years)
Decline in Panama functional class | Over registry run-time (5.5 years)
Worsening of echocardiographic parameters (ECHO) | Over registry run-time (5.5 years)
  Parameters encompass TAPSE and RV/LV dimension ratio
Increase in Brain Natriuretic Peptide (BNP) | Over registry run-time (5.5 years)
Increase in N-terminal-proBNP (NT-proBNP) | Over registry run-time (5.5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Dunbar Ivy, Prof, Study Chair — Association for Pediatric Pulmonary Hypertension
Locations (32):
- United States (13):
  - Stanford Children's Hospital, Palo Alto, California
  - University of Colorado Denver School of Medicine, Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - St Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University Children's Hospital, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Royal Children's Hospital, Melbourne, Australia
- University of São Paulo, São Paulo, Brazil
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Fu Wai Hospital, Beijing, China
- Hospital Pediátrico La Misericordia, Bogotá, Colombia
- Université Paris Descartes, Paris, France
- University Children's Hospital Ulm, Ulm, Germany
- Institute of Cardiology, Budapest, Hungary
- Hadassah, Hebrew University Medical Center, Jerusalem, Israel
- University of Padova, Padua, Italy
- Japan (2):
  - Toho Universit Omori Medical Center, Tokyo
  - Keio University, Tokyo
- National Heart Institute, Mexico City, Mexico
- Beatrix Children's Hospital, University Medical Center Groningen, Groningen, Netherlands
- Children's Memorial, Warsaw, Poland
- King Fahd Armed Forces Hospital, Jeddah, Saudi Arabia
- The Queen Silvia's Children's Hospital, Gothenburg, Sweden
- Switzerland (2):
  - Hôpital des Enfants, Geneva
  - University Children's Hospital, Zurich

REFERENCES:
- See also: Webpage of the Association for Pediatric Pulmonary Hypertension — https://www.peph-association.org/